CLINICAL TRIAL: NCT06831253
Title: Efficacy of Restoration of Lacrimal Secretion After Injection of Platelet-Rich Plasma (PRP) Into the Lacrimal Gland in Severe Dry Eye Syndromes (ReLIPSSO)
Brief Title: Efficacy of Platelet-Rich Plasma Injection in Dry Eye Syndrome
Acronym: ReLIPSSO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-AOIP-02; IDRCB (Other: 2024-A02096-41)
Record Dates: First submitted 2025-02-07; First posted 2025-02-18 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Severe Dry Eye Syndromes; Dry Eye Syndromes
Keywords: Dry Eye Syndromes; lacrimal gland; platelet-rich plasma; aqueuous deficiency
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Masking Description: To assess the lacrimal secretion after 4 injections of PRP in lacrimal gland
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Injection of Platelet-Rich Plasma (PRP) (Experimental)
  Interventions: Other: injections of Platelet-Rich Plasma in lacrimal gland

INTERVENTIONS:
Other: injections of Platelet-Rich Plasma in lacrimal gland — injections of Platelet-Rich Plasma in lacrimal gland

SUMMARY:
The investigatror wants to show the efficacy of Platelet-Rich Plasma injection in lacrimal gland to restore the lacrimal secretion in patients presenting aqueous deficiency reponsible for severe dry eye syndrome.

DETAILED DESCRIPTION:
injections in lacrimal gland four times during the study for each patient

ELIGIBILITY:
Inclusion Criteria:

* Platelet counts, and clotting factors in the standarts
* Presenting with severe dry keratoconjunctivitis diagnosed by an ophthalmologist

Exclusion Criteria:

* Patients with significant fibrosis of the conjunctival portion of the lacrimal gland
* Patients with complete stenosis of both lacrimal meatus in the treated eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
To compare the lacrimal secretion after 4 monthly injections of PRP into the lacrimal gland | week 16
  Schirmer I test score between 0mm and more 20mm

SECONDARY OUTCOMES:
To compare the different clinical follow-up parameters of qualitative dry ocular syndrome and quantitative after 4 monthly injections of PRP into the lacrimal gland | week 16
  Ocular Surface Diseases Index (OSDI) a scale of 0 to 100

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, Site Principal Investigator, France

IPD SHARING:
Plan to Share IPD: No